CLINICAL TRIAL: NCT00611897
Title: N-acetylcysteine and NMDA Antagonist Interactions
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple
Other Study IDs: 0508000518
Record Dates: First submitted 2008-01-29; First posted 2008-02-11 (Estimated); Results first posted 2015-05-08 (Estimated); Last update posted 2015-05-08 (Estimated); Status verified 2015-05

CONDITIONS: Cognitive Dysfunction
Keywords: NMDA; glutamate; N-acetylcysteine; P3
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Acetylcysteine; Ketamine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (Active Comparator): The NAC capsules were administered orally in divided doses: 2000 mg followed by 1000 mg 2 hours later. Each morning, 165 min after NAC administration, subjects received a 1-min bolus of normal saline, followed by a 70-minlong saline infusion during which behavioral, cognitive, and ERP data were collected. Ketamine was administered intravenously as a bolus of .23 mg/kg over 1 min followed by .58 mg/kg for 30 min (SPM and RVP), and then .29 mg/kg for 40 min (P300 and MMN).
  Interventions: Drug: N-acetylcysteine and ketamine
- Arm II (Placebo Comparator): The placebo capsules were administered orally in divided doses: 2000 mg followed by 1000 mg 2 hours later. Each morning, 165 min after placebo administration, subjects received a 1-min bolus of normal saline, followed by a 70-minlong saline infusion during which behavioral, cognitive, and ERP data were collected. Ketamine was administered intravenously as a bolus of .23 mg/kg over 1 min followed by .58 mg/kg for 30 min (SPM and RVP), and then .29 mg/kg for 40 min (P300 and MMN).
  Interventions: Drug: placebo and ketamine

INTERVENTIONS:
Drug: N-acetylcysteine and ketamine — Active drug (N-acetylcysteine)
  Other Names: NAC
  Arms: Arm I
Drug: placebo and ketamine — placebo N-acetylcysteine
  Arms: Arm II

SUMMARY:
This study tests the hypothesis that extrasynaptic mechanisms are critically linked with cognitive effects of NMDA antagonism as evidenced by event-related potentials (ERPs) in healthy humans.

ELIGIBILITY:
Inclusion Criteria:

* Ages of 21-45 years from all ethnic backgrounds.
* Male or female.
* Written informed consent.

Exclusion criteria

* DSM-IV diagnosis for a psychotic, depressive or anxiety disorder.
* A history of significant medical/neurological disease such as cardiac, thyroid, renal, hepatic abnormality, seizure disorder. Unstable medical condition based on EKG, vital signs, physical examination and laboratory work-up (CBC with differential, SMA-7, LFTs, TFTs, UA, Utox, Urine pregnancy test) .
* History of severe allergies or multiple adverse drug reactions.
* Any medication that in the opinion of the PI could interfere with either the safety of the study and/or the outcome measures.
* Any other conditions which in the opinion of the investigator would preclude participation in the study.
* History of major psychiatric disorder in first degree relatives.
* Current substance abuse/dependency determined by urine toxicology.
* Current treatment with medications with psychotropic effects.
* Treatment with benzodiazepines within one week prior to testing.
* Current pregnancy, unsatisfactory birth control method report for females.
* Education < 10th grade.
* IQ < 70, MR as determined by Wechsler Abbreviated Scale of Intelligence.
* Non-English speaking.

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2006-01; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Handan Gunduz-Bruce, M.D., Principal Investigator — Yale University
Locations (1):
- VHA Connecticut, West Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was approved by the institutional review boards of Yale Medical School and the Veterans Administration Connecticut Healthcare System. Healthy volunteers were recruited by advertisements.
  as determined by Structured Clinical Interview for DSM-IV, Non-Patient Edition.
Pre-assignment Details: All subjects gave written informed consent. They had no personal or family history of psychiatric or substance abuse disorders. A total of 43 subjects consented; 21 of them never initiated the study due to ineligibility or scheduling conflicts, and 6 subjects dropped out. Sixteen subjects completed the study procedures.
Groups:
- Day 1: Active NAC; Day 2: Placebo NAC: Subjects were randomized to receive ACTIVE NAC on day one, before the infusion of saline and then ketamine (as a bolus of .23 mg/kg over 1 min followed by .58 mg/kg for 30 min, and then .29 mg/kg for 40 min) in a fixed order. Subjects then received PLACEBO NAC on day two, before the infusion of saline and then ketamine (as a bolus of .23 mg/kg over 1 min followed by .58 mg/kg for 30 min, and then .29 mg/kg for 40 min) in a fixed order.
- Day 1: Placebo NAC; Day 2: Active NAC: Subjects were randomized to receive PLACEBO NAC on day one, before the infusion of saline and then ketamine (as a bolus of .23 mg/kg over 1 min followed by .58 mg/kg for 30 min, and then .29 mg/kg for 40 min) in a fixed order. Subjects then received ACTIVE NAC on day two, before the infusion of saline and then ketamine (as a bolus of .23 mg/kg over 1 min followed by .58 mg/kg for 30 min, and then .29 mg/kg for 40 min) in a fixed order.
Period: Day 1: Initial Treatment
Arm/Group | Day 1: Active NAC; Day 2: Placebo NAC | Day 1: Placebo NAC; Day 2: Active NAC
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0
Period: Day 2: Crossover Treatment
Arm/Group | Day 1: Active NAC; Day 2: Placebo NAC | Day 1: Placebo NAC; Day 2: Active NAC
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Sample: This is the group of healthy volunteers that consented to participate in the study.
Arm/Group | Overall Sample
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.0 (5.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 13

OUTCOME MEASURES:

1. Primary Outcome: Target P300
Description: The Target P300 measures were obtained from the Fz, Cz and Pz electrodes.
  Target stimuli were 1000 Hz tones (500 ms) and novel stimuli (~250 ms) were unique environmental sounds (e.g., dog bark) used in prior studies of the novelty P300. Subjects were instructed to respond to the target sounds by pressing a button using their dominant hand index finger. The standard stimuli were 20, 30 or 40 Hz click trains (500 ms) in the first, second, and third runs, respectively. The auditory steady state EEG driving data obtained from these standard stimuli will be presented in a separate report. All stimuli were presented at 80 dB SPL.
Time Frame: daily
Population: Per protocol
Measure: Least Squares Mean (Standard Error); unit: microvolts
Groups:
- Placebo+Saline: NAC placebo capsule administered after receiving 1-min bolus of saline, followed by a 70-min long saline infusion during which behavioral, cognitive, and ERP data were collected.
- Placebo+Ketamine: NAC placebo capsule, Ketamine was administered intravenously as a bolus of .29 mg/kg for 40 min.
- NAC+Saline: NAC active capsule administered after receiving 1-min bolus of saline, followed by a 70-min long saline infusion during which behavioral, cognitive, and ERP data were collected.
- NAC+Ketamine: NAC active capsule, Ketamine was administered intravenously as a bolus of .29 mg/kg for 40 min.
Arm/Group | Placebo+Saline | Placebo+Ketamine | NAC+Saline | NAC+Ketamine
Number analyzed (Participants) | 16 | 16 | 16 | 16
microvolts
  Fz | 2.5 (0.8) | 3.2 (0.8) | 5.2 (0.8) | 3.4 (0.8)
  Cz | 7.7 (1.0) | 5.5 (1.0) | 9.9 (1.0) | 5.4 (1.0)
  Pz | 11.8 (1.1) | 8.1 (1.1) | 12.6 (1.1) | 8.2 (1.1)

2. Secondary Outcome: Mismatch Negativity (MMN) Intensity
Description: Mismatch Negativity (MMN) Intensity difference waves at midline electrodes (Fz, Cz and Pz).
  The frequent standard tones were of 75 ms duration with 5 ms rise and fall time, and were composed of 500, 1000, and 1500 Hz sinusoidal partials (harmonics) that resulted in a single high pitched beep sound.
  All tones were presented at 76 dB sound pressure level (SPL) with the exception of intensity deviants. The three deviants were distinguishable from standard tones in either intensity, frequency, or duration.
  Subjects performed a visual discrimination distractor task during the MMN runs and were instructed to ignore the tones.
  The mismatch negativity (MMN) measure included 3 types of deviant tones (stimuli) that the subjects heard: 1. Frequency deviant, 2. Intensity deviant, 3. Duration deviant. The response to these 3 types of deviants were recorded in the EEG. Therefore each deviant was associated with different waves which we measured in amplitude (microvolts)
Time Frame: daily
Population: Per protocol
Measure: Least Squares Mean (Standard Error); unit: microvolts
Arm/Group | Placebo+Saline | Placebo+Ketamine | NAC+Saline | NAC+Ketamine
Number analyzed (Participants) | 16 | 16 | 16 | 16
microvolts
  Fz | -3.5 (0.2) | -2.7 (0.2) | -3.4 (0.2) | -2.6 (0.2)
  Cz | -3.2 (0.2) | -2.5 (0.2) | -3.4 (0.2) | -2.6 (0.2)
  Pz | -2.1 (0.2) | -2.0 (0.2) | -2.4 (0.2) | -2.1 (0.2)

3. Primary Outcome: Novel P300
Description: The Novel P300 measures were obtained from the Fz, Cz and Pz electrodes.
  Target stimuli were 1000 Hz tones (500 ms) and novel stimuli (~250 ms) were unique environmental sounds (e.g., dog bark) used in prior studies of the novelty P300. Subjects were instructed to respond to the target sounds by pressing a button using their dominant hand index finger. The standard stimuli were 20, 30 or 40 Hz click trains (500 ms) in the first, second, and third runs, respectively. The auditory steady state EEG driving data obtained from these standard stimuli will be presented in a separate report. All stimuli were presented at 80 dB SPL.
Time Frame: daily
Population: Per protocol
Measure: Least Squares Mean (Standard Error); unit: microvolts
Arm/Group | Placebo+Saline | Placebo+Ketamine | NAC+Saline | NAC+Ketamine
Number analyzed (Participants) | 16 | 16 | 16 | 16
microvolts
  Fz | 5.6 (0.8) | 5.2 (0.8) | 7.6 (0.8) | 5.3 (0.8)
  Cz | 10.5 (1.0) | 7.0 (1.0) | 11.5 (1.0) | 7.4 (1.0)
  Pz | 10.7 (1.2) | 5.7 (1.2) | 10.8 (1.2) | 6.1 (1.2)

4. Secondary Outcome: Mismatch Negativity (MMN) Frequency
Description: Mismatch Negativity (MMN) Frequency difference waves at midline electrodes (Fx, Cz and Pz).
  The frequent standard tones were of 75 ms duration with 5 ms rise and fall time, and were composed of 500, 1000, and 1500 Hz sinusoidal partials (harmonics) that resulted in a single high pitched beep sound.
  All tones were presented at 76 dB sound pressure level (SPL) with the exception of intensity deviants. The three deviants were distinguishable from standard tones in either intensity, frequency, or duration.
  Subjects performed a visual discrimination distractor task during the MMN runs and were instructed to ignore the tones.
  The mismatch negativity (MMN) measure included 3 types of deviant tones (stimuli) that the subjects heard: 1. Frequency deviant, 2. Intensity deviant, 3. Duration deviant. The response to these 3 types of deviants were recorded in the EEG. Therefore each deviant was associated with different waves which we measured in amplitude (microvolts)
Time Frame: daily
Population: Per protocol
Measure: Least Squares Mean (Standard Error); unit: microvolts
Arm/Group | Placebo+Saline | Placebo+Ketamine | NAC+Saline | NAC+Ketamine
Number analyzed (Participants) | 16 | 16 | 16 | 16
microvolts
  Fz | -3.3 (0.3) | -2.7 (0.3) | -3.1 (0.2) | -2.9 (0.2)
  Cz | -3.3 (0.3) | -2.7 (0.3) | -3.1 (0.2) | -2.9 (0.2)
  Pz | -2.3 (0.2) | -1.7 (0.2) | -1.8 (0.2) | -1.9 (0.2)

5. Secondary Outcome: Mismatch Negativity (MMN) Duration
Description: Mismatch Negativity (MMN) Duration difference waves at midline electrodes (Fz, Cz and Pz).
  The frequent standard tones were of 75 ms duration with 5 ms rise and fall time, and were composed of 500, 1000, and 1500 Hz sinusoidal partials (harmonics) that resulted in a single high pitched beep sound.
  All tones were presented at 76 dB sound pressure level (SPL) with the exception of intensity deviants. The three deviants were distinguishable from standard tones in either intensity, frequency, or duration.
  Subjects performed a visual discrimination distractor task during the MMN runs and were instructed to ignore the tones.
  The mismatch negativity (MMN) measure included 3 types of deviant tones (stimuli) that the subjects heard: 1. Frequency deviant, 2. Intensity deviant, 3. Duration deviant. The response to these 3 types of deviants were recorded in the EEG. Therefore each deviant was associated with different waves which we measured in amplitude (microvolts)
Time Frame: daily
Population: Per protocol
Measure: Least Squares Mean (Standard Error); unit: microvolts
Arm/Group | Placebo+Saline | Placebo+Ketamine | NAC+Saline | NAC+Ketamine
Number analyzed (Participants) | 16 | 16 | 16 | 16
microvolts
  Fz | -3.2 (0.3) | -3.1 (0.3) | -3.2 (0.3) | -2.8 (0.3)
  Cz | -3.1 (0.3) | -3.1 (0.3) | -3.3 (0.3) | -2.8 (0.3)
  Pz | -2.4 (0.2) | -2.3 (0.2) | -2.4 (0.2) | -2.1 (0.2)

ADVERSE EVENTS:
Time Frame: Adverse events were collected across the duration of the intervention in both arms. These data were not collected at the specific intervals in either arm.
Arm/Group | Day 1: Placebo NAC; Day 2: Active NAC | Day 1: Active NAC; Day 2: Placebo NAC
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 4/8 | 0/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Day 1: Placebo NAC; Day 2: Active NAC (N=8) | Day 1: Active NAC; Day 2: Placebo NAC (N=8)
Nausea (Gastrointestinal disorders) | 4 (4) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes